CLINICAL TRIAL: NCT06030544
Title: Oleanolic Acid as Therapeutic Adjuvant for Type 2 Diabetes Mellitus (OLTRAD STUDY)
Acronym: OLTRAD
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish National Research Council (Other Government)
Collaborators: Andalusian Health Service (Other Government); Universidad Pablo de Olavide (Other)
Responsible Party: Principal Investigator, José M. Castellano, PhD, Principal Investigator, Spanish National Research Council
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PID2019-107837RB-I00
Record Dates: First submitted 2023-07-24; First posted 2023-09-11 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Diabetic Patients; Type II Diabetes Mellitus
Keywords: Oleanolic acid; T2DM treatment; randomized controlled trial; parallel groups design; dietary intervention; functional olive oil
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Oleanolic Acid

STUDY DESIGN:
Intervention Model Description: prospective, parallel group, randomized, double-blind, controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both the OA-enriched olive oil and the control oil will be delivered labeled with alphanumeric codes, the correspondence of which will only be known by the Dr. Jose M. Castellano (Principal Investigator 1). This ensures blinding of the other researchers and trial participants with respect to the type of olive oil assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OA-enriched functional olive oil (Experimental): Functional olive oil elaborated enriching the control olive oil with high purity (> 95 %) Oleanolic acid from olive leaf up to 600 mg OA/kg oil.
  Interventions: Dietary Supplement: OA-enriched functional olive oil
- Control olive oil (Active Comparator): Commercial olive oil (blend of virgin and refined olive oils) chosen by its very low content of bioactive minor components.
  Interventions: Dietary Supplement: commercial olive oil

INTERVENTIONS:
Dietary Supplement: OA-enriched functional olive oil — Dietary intervention in diabetic patients. Oral intake of 55 mL/day of a functional olive oil enriched in Oleanolic acid (equivalent dose 30 mg/day OA) Oleanolic acid (CAS no. 598-02-1; PubChem CID 10494).
  Other Names: Functional olive oil enriched in Oleanolic acid
  Arms: OA-enriched functional olive oil
Dietary Supplement: commercial olive oil — Dietary intervention in diabetic patients. Oral intake of 55 mL/day of a commercial olive oil (blend of virgin and refined olive oils) chosen by its very low content of bioactive minor components.
  Other Names: control olive oil
  Arms: Control olive oil

SUMMARY:
Oleanolic acid (OA), is a natural component of many plant food and medicinal herbs, which has shown to exert in experimental models hypoglycemic and hypolipidemic effects, and also a cytoprotective action against oxidative and chemotoxic stress underlying Type II Diabetes Mellitus (T2DM).Today it is known that OA shares mechanisms of action with metformin and other drugs of choice for the treatment of diabetes. Therefore, the OLTRAD (OLeanolic acid TReAtment for type 2 Diabetes) Study, a prospective, parallel group, randomized, double-blind, controlled trial with 100 participants, has been designed to demonstrate that the regular intake of an OA-enriched functional olive oil is effective as an adjuvant to metformin antidiabetic drug therapy. The hypothesis is that the inclusion of this functional olive oil in the diet will enhance the effects of the pharmacological treatment in diabetic patients, and may even reduce the need for prescription of such medications.

DETAILED DESCRIPTION:
TRIAL DESIGN The OLTRAD Study is a prospective, parallel group, randomized, double-blind, controlled trial designed to demonstrate that the regular intake of an OA-enriched functional olive oil is effective as an adjunct to metformin therapy (as monotherapy or in combination with other antidiabetic drugs) in the metabolic control of T2DM patients. The effect of the OA-enriched olive oil will be compared with that of the control oil, which consists of the same commercial olive oil not fortified in the triterpene.

A total of 100 volunteers of both sex will be selected from among the T2DM patients treated at the Endocrinology and Nutrition Service of the 'Virgen del Rocío' University Hospital (Seville, SPAIN).

SAMPLE SIZE CALCULATION Serum glycosylated hemoglobin (HbA1c) is adopted as the main quantitative variable for the analysis of glycemic control. The null hypothesis stated in the trial design is that the OA-based dietary intervention will reduce the baseline serum HbA1c levels of patients by at least 7%, compared to the control group. To test this one-sided hypothesis test with a 95% confidence level (α risk = 0.05) and 95% power (β risk = 0.05), a sample size of 44 volunteers per group is required. However, due to the characteristics of the study (a long-term lifestyle intervention), participant losses of up to 15% can be assumed, resulting in an adjusted sample size of 50 individuals per group.

RANDOMIZATION Once recruited, the 100 T2DM patients will be randomly assigned to one of the two study groups. Fifty individuals will be assigned to the intervention group, which will ingest the OA-enriched functional olive oil, whereas the other 50 volunteers will be assigned to the control group, which will receive the same non-enriched olive oil. At the time of admission, the study nursing staff will request by telephone the clinical coordinator of the trial (Principal Investigator 2 of the Project) the assignment of participants to the study groups (centralized randomization). Allocation to these groups will be made using computer generated tables of random numbers. Four randomization strata will be constructed by sex and age (cuttof 50 years).

INTERVENTION Participants will be instructed to ingest 55 mL/day of the assigned oil, preferably raw and freely distributed among the three main meals. Both the OA-enriched olive oil and the control oil will be delivered labeled with alphanumeric codes, the correspondence of which will only be known by the Principal Investigator 1 of the project. This ensures blinding of the clinical researchers and participants with respect to the type of olive oil assigned.

FOLLOW-UP Participants in the clinical trial will be followed up for 12 months from enrollment, according to a plan of quarterly visits.

At the time of recruitment and every three months thereafter, participants will be measured for anthropometric, blood pressure, and heart rate measurements. They will also be asked about gastrointestinal disorders or other types of complaints, and will complete a questionnaire on lifestyle (diet, physical activity, alcohol and tobacco use), medical conditions, and medication use.

Also at the beginning of participation in the study and every three months thereafter, fasting blood samples will be drawn from the cubital vein, which will be collected in sterile plastic tubes with a vacuum system. Similarly, participants will provide aliquots of their first morning urine in sterile plastic tubes. The analytical determinations in blood and urine will be carried out in the Clinical Biochemistry and Analysis Laboratory of the 'Virgen del Rocío' University Hospital in Seville (HUVR).

In addition, aliquots of plasma will be sent to the 'Instituto de la Grasa' (IG-CSIC) for complementary biochemical determinations. Laboratory technicians from both institutions will receive the samples identified with alphanumeric ID codes and, therefore, will be blinded to the intervention groups.

In these quarterly visits, volunteers will participate in sessions of the nutritional education program and will receive 6 L of the assigned oil for free. Adherence to the dietary intervention will be assessed quarterly through the Haynes-Sackett's self-reported compliance test and the return of empty bottles presumably consumed.

The primary outcome of the trial is the improvement in glycemic control, assessed by the evolution of HbA1c. As secondary results, we will obtain data on anthropometric and clinical variables, as well as on biochemical parameters of blood and urine.

ANAMNESIS AND CLINICAL EXAMINATION OF PARTICIPANTS The medical researchers of the project have access to the electronic medical records of the participants in the platform DIRAYA of the Andalusian Health Service, and will carry out the anamnesis and physical examination of the participants, which will include vital data and general medical and surgical history, as well as the pharmacological treatments followed. Information will also be obtained on lifestyle, perception of their own body image, diet, and the type and intensity of physical activity. In addition, a general clinical examination will be carried out including general appearance and inspection of hands and arms, feet and legs, skin, face, eyes, mouth, neck, abdomen, edema, lymph nodes, and vital signs (temperature, pulse, respiratory rate and blood pressure).

ANTHROPOMETRIC STUDY AND BODY COMPOSITION The anthropometric study will include the determination of total body weight, height, body mass index (BMI), as well as waist and hip circumferences. The study and evaluation of these variables will be carried out according to the guidelines of the International Society for the Advancement of Kinanthropometry (ISAK). The study of body composition will be carried out by electrical bioimpedance. Fat mass, lean mass, muscle mass, total water, bone mass, basal metabolism, and visceral fat will be quantified with this technique, using validated prediction equations adjusted for age and sex.

ASSESSMENT OF FOOD INTAKE AND NUTRITIONAL TRAINING A nutritional education program will be implemented to assess the food intake of the participants and reinforce compliance with the dietary recommendations given. To measure food intake, we will use the food intake registration form designed by the University of Navarra (Spain) and used successfully in other trials, such as the PREvención con DIeta MEDiterránea (PREDIMED) study. This form is a validated tool that quantifies food intake in terms of food portions or food groups for adults living in Spain. On the other hand, all the participants will join workshops where they will receive specific dietary recommendations for patients with T2DM, and they will be instructed on a healthy diet, the best food options and adequate portions, limiting highly processed foods, cakes, sugar, fatty foods as well as sugary and alcoholic beverages. Additionally, patients will gain information on recipes, seasonal shopping lists, and the use of olive oil for cooking and dressing. The eating habits of the participants will be analyzed quarterly by means of a 24-hour recall questionnaire. The 'NUTRIUM' software (https://nutrium.com/; Braga; Portugal) for the nutritional evaluation of the diets will be used.

BLOOD BIOCHEMISTRY IN HUVR In ulnar blood samples, determinations related to circulating lipids [total triglycerides, total cholesterol, LDL, HDL, total apolipoprotein B and lipoprotein A]; glucose homeostasis [glycemia, insulinemia, C-peptide, HOMA-IR index, HbA1c]; oxidative stress and inflammation [uric acid, bilirubin, malondialdehyde, ultrasensitive C-reactive protein, thyroid-stimulating hormone (TSH)], as well as those associated with liver and kidney damage [lactate dehydrogenase (LDH), liver transaminases (ALT, AST, GGT ) and creatinine] will be performed.

Plasma level of vitamin B12 will be also assessed. In addition, the possible appearance of liver fibrosis will be evaluated through the Hepamet Fibrosis Score, a non-invasive method that calculates a score taking into account factors such as age, sex, presence of diabetes, glucose levels, insulin, albumin, platelets, and AST. This tool, designed by the Seville Institute of Biomedicine (IBiS), is indicated to assess suspected fibrosis in patients with obesity, diabetes, metabolic syndrome, hepatic steatosis, and/or abnormal liver function markers. The method offers diagnostic reliability and a cost/benefit ratio that is superior to other methods, such as the FIB-4 and the NAFLD Fibrosis Score.

CONTINUOUS BLOOD GLUCOSE MONITORING Plasma glucose will be continuously monitored using the 'FreeStyle Libre' subcutaneous system (ABBOTT Diagnostics; Chicago, IL.; USA). The sensors will be attached to the participants at two times throughout the trial: at baseline and after 12 months of follow-up, and will collect data for 48 hours. With this system, different glycemic parameters will be determined, such as the area under the curve (AUC), the mean amplitude of the glycemic excursion (MAGE), the mean glycemia, as well as the standard deviation (SD) and the coefficient of variation (CV).

PLASMA BIOCHEMISTRY IN IG-CSIC The investigators of the IG-CSIC will perform a number of complementary determinations in plasma samples, such as the plasmatic concentrations of OA, the glutathione (GSH and GSSG) levels, the fatty acid composition, serum adipokines (ceruloplasmin, adiponectin, leptin, resistin, and ghrelin). Serum Antioxidant enzymes (superoxide dismutase, catalase) and proinflammatory cytokines (TNF-α, IL-1β, IL-6) will also be determined.

On the other hand, the VLDL fraction of plasma lipoproteins will be isolated by ultracentrifugation (230,000 × g for 18 h at 4 °C). In these particles, the total content of fatty acids, triglycerides, diglycerides, phospholipids and total Apolipoprotein B will be measured.

URINE ANALYSIS The first morning urine samples will be analyzed for the usual physical, chemical, and microscopic determinations (pH, density, glycosuria, ketones, nitrites, urobilinogen, bilirubin, sediment, leukocytes, microalbuminuria/g creatinine). The determination of these parameters will also be carried out in the facilities of the Clinical Biochemistry and Analysis Laboratory of the 'Virgen del Rocío' University Hospitals in Seville.

STATISTICAL ANALYSIS The trial will be conducted according to the intention-to-treat (ITT) principle. Qualitative variables will be expressed by their absolute and relative frequencies, whereas the quantitative ones with normal distribution will be expressed by the mean and standard deviation and those with non-normal distribution by the median and interquartile range (IQR). Comparisons between study groups for qualitative variables will be performed with the Chi-square and McNemar's tests, whereas comparisons for quantitative variables will be executed with the Student's t-test and ANOVA. The homogeneity of the populations included in the allocation groups will be evaluated using theMann-Whitney-Wilcoxon U-test. All P-values will be two-tailed at α = 0.05. Statistical analysis will be performed with SPSS 27 (IBM SPSS Statistics, NY, USA) software

ELIGIBILITY:
Inclusion Criteria:

1. community-residing men and women aged.
2. Body Mass Index (BMI) between 25 and 39.9 kg/m2.
3. diagnosed with T2DM [Following the American Diabetes Association (ADA) 2019 criteria] at least six months before being included in this trial.
4. be treated with metformin (stable dose >= 850 mg/day at least three months before recruitment) as monotherapy, or in combination with other hypoglycemic agents (administration of insulin exclusively in a single basal dose), except pioglitazone and sulphonylureas.
5. HbA1c below 9% at baseline, with a variation compared with a prior HbA1c from at least three months before inclusion in this trial of less than +/- 0.5 %.
6. be able to give voluntary informed consent and willing to comply with all study procedures.

Exclusion Criteria:

1. suffering from Type 1 Diabetes Mellitus or latent autoimmune diabetes in adults.
2. suffering from chronic kidney disease (estimated glomerular filtration rate (eGFR) <30 ml/min/1.73m2).
3. suffering from acute or chronic hepatitis, signs and symptoms of any liver disease other than non-alcoholic fatty liver disease (NAFLD), or ALT/AST ratio >3 times the upper limit of the reference range.
4. To present, at the time of recruitment, allergies and intolerances associated with food consumption.
5. pregnant and lactating women.
6. lack of willingness to use a highly effective contraceptive method (in women of childbearing potential).
7. fasting triglyceridemia > 600 mg/dL despite adequate treatment.
8. grade 3 hypertension (systolic blood pressure ≥ 180 mm Hg and/or diastolic blood pressure ≥ 110 mm Hg) according to the 2018 guidelines of the European Society of Hypertension.
9. use of pioglitazone or sulfonylureas.
10. being treated with medications that promote weight loss (eg, Saxenda® [liraglutide 3.0 mg], Xenical® [orlistat], or similar over-the-counter [OTC] medications) within six months prior to the start of the trial.
11. Being on chronic (>14 days) therapy with systemic glucocorticoids (excluding topical, intraocular, intranasal, intra-articular, or inhaled preparations) within six months prior to enrollment.
12. Presenting any of the following cardiovascular conditions within 6 months prior to study entry: acute myocardial infarction, unstable angina, New York Heart Association (NYHA) class III or class IV heart failure, or cerebrovascular accident.
13. Evidence, in the investigators' opinion, of significant uncontrolled endocrine abnormality (e.g., thyrotoxicosis, adrenal crisis) at baseline.
14. History of active or untreated malignancy, or being in remission from a clinically significant malignancy (other than basal or squamous cell skin cancer, cervical carcinoma in situ, or prostate cancer in situ) during the last 5 years before the study entry.
15. Participation in the last 30 days in a clinical trial with an investigational product [if the previous investigational product has a long half-life, 3 months or 5 half-lives (whichever is longer) should have passed].
16. Being, at the time of recruitment, enrolled in any other clinical trial involving an investigational product or any other type of medical research that is not considered scientifically or medically compatible with this study.
17. Presence of any hematologic condition that may interfere with HbA1c measurement (eg, hemolytic anemias, sickle cell anemia).
18. History of any other condition (eg, known drug or alcohol abuse or psychiatric disorder, or any other physical or intellectual limitations), which, in the opinion of the investigator, may prevent the patient from following and completing the protocols.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-02-25 (Actual); Primary Completion 2025-03-20 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 1 year
  The primary outcome of the trial is the evaluation of the glycemic control, assessed through the evolution of the plasma glycosylated hemoglobin (HbA1c) level, expressed in %

SECONDARY OUTCOMES:
Body weight | 1 year
  Body weight (expressed in kilograms, kg) wil be determined using a TANITA® model BC-418MA body composition analyzer.
Body height | 1 year
  The body height (expressed in meters, m) will be determined by using an approved column stadiometer
Body mass index (BMI) | 1 year
  body weight and height will be combined to report BMI in kg/m^2, according to the equation BMI = body mass/(height)^2
Waist circumference | 1 year
  Waist circumference (expressed in centimeters, cm) will be measured with a measuring tape
Hip circumference | 1 year
  Hip circumference (expressed in centimeters, cm) will be measured with a measuring tape
Body composition - fat mass | 1 year
  Fat mass (expressed in kilograms, kg) will be measured using a TANITA® (model BC-418MA) body composition analyzer. Quantification will be made using validated prediction equations adjusted for age and sex.
Body composition - visceral fat mass | 1 year
  Visceral fat mass (expressed in kilograms, kg) will be measured using a TANITA® (model BC-418MA) body composition analyzer. Quantification will be made using validated prediction equations adjusted for age and sex.
Body composition - lean mass | 1 year
  Lean mass (expressed in kilograms, kg) will be measured using a TANITA® (model BC-418MA) body composition analyzer. Quantification will be made using validated prediction equations adjusted for age and sex.
Body composition - muscle mass | 1 year
  Muscle mass (expressed in kilograms, kg) will be measured using a TANITA® (model BC-418MA) body composition analyzer. Quantification will be made using validated prediction equations adjusted for age and sex.
Body composition - bone mass | 1 year
  Bone mass (expressed in kilograms, kg) will be measured using a TANITA® (model BC-418MA) body composition analyzer. Quantification will be made using validated prediction equations adjusted for age and sex.
Body composition - total water composition | 1 year
  Total water composition (expressed in litre, L) will be measured using a TANITA® (model BC-418MA) body composition analyzer. Quantification will be made using validated prediction equations adjusted for age and sex.
Basal metabolism | 1 year
  Basal metabolism (expressed in kilojoule, kJ) will be measured using a TANITA® (model BC-418MA) body composition analyzer. Quantification will be made using validated prediction equations adjusted for age and sex.
Diastolic blood pressure (DBP) | 1 year
  DBP (expressed in milimeters of mercury) using a calibrated automatic sphygmomanometer
Systolic blood pressure (SBP) | 1 year
  SBP (expressed in milimeters of mercury) using a calibrated automatic sphygmomanometer
Pulse | 1 year
  heart rate measured with a calibrated automatic sphygmomanometer
Serum glucose | 1 year
  Determined by enzymatic method and expressed in miligrams/decilitre (mg/dL)
Serum insulin | 1 year
  determined by commercial ELISA kit and expressed in international microunits per millilitre (µIU/mL)
HOMA-IR index | 1 year
  serum glucose (expressed in millimole/litre) and serum insulin (expressed in µIU/mL) are combined to report the homeostatic model assessment for insulin resistance (HOMA-IR), according to the equation HOMA-IR = (glucose x insulin)/22.5 HOMA-IR= [serum insulin (μU/ml) × blood glucose (mmol/l)]/22.5}.
Serum C-peptide | 1 year
  measured by commercial ELISA kit and expressed as nanogram/millilitre (ng/mL)
Plasma triglycerides (TG) | 1 year
  plasma concentrations of total triglycerides is determined by an automated colorimetric enzymatic method (GPO-PAP, Roche Diagnostics, Mannheim, Germany) and expressed as milligrams/decilitre (mg/dL)
Plasma total cholesterol (CT) | 1 year
  plasma concentrations of total cholesterol is determined by an automated colorimetric enzymatic method (CHOD-PAP, Roche Diagnostics, Mannheim, Germany) and expressed as milligrams/decilitre (mg/dL)
Plasma high density lipoproteins (HDL) | 1 year
  plasma concentrations of HDL is determined by an automated direct enzymatic method (HDL-C-plus 2nd generation, Roche Diagnostics, Mannheim, Germany) and expressed as milligrams/decilitre (mg/dL)
Plasma low density lipoproteins (LDL) | 1 year
  Triglycerides, total cholesterol and high densitity lipoproteins are combined to report LDL, according to the Friedewald formula:
  LDL = CT - (TG/ 5) - HDL
Plasma lipoprotein A | 1 year
  the plasma content of lipoprotein A is quantified by ELISA and the values are expressed as milligram/decilitre (mg/dL)
Plasma total lipoprotein B | 1 year
  the plasma content of total lipoprotein B (Apo B48 + Apo B100) is quantified by an immunoturbidimetric assay (Tinaquant; Roche Diagnostics, Mannheim, Germany), The values are expressed as milligram/decilitre (mg/dL)
Plasma creatinine | 1 year
  standard spectrophotometric assay. Values expressed as milligrams per decilitre (mg/dL)
Plasma uric acid | 1 year
  Evaluated by an enzymatic procedure, with results expressed in milligrams per decilitre (mg/dL)
Plasma alanine aminotransferase (ALT) | 1 year
  use of a diagnose kit with values expressed as units per litre (U/L)
Plasma aspartate aminotransferase (AST) | 1 year
  use of a diagnose kit with values expressed as units per litre (U/L)
Plasma gamma-glutamyl transferase (GGT) | 1 year
  use of a diagnose kit with values expressed as units per litre (U/L)
Plasma lactate dehydrogenase (LDH) | 1 year
  L-Lactic Dehydrogenase kit. Results expressed as units per litre (U/L)
Plasma bilirubin | 1 year
  Spectrofotometric assay. Results expressed as milligrams per decilitre (mg/dL)
Plasma levels of glutathion (GSH and GSSG) | 1 year
  Glutathione Reductase (GR) Assay Kit. Values expressed as milliunits per millilitre (mU/mL)
Plasma malondialdehyde | 1 year
  Thiobarbituric acid (TBA) assay and HPLC determination. Results expressed as µmole per litre (µmol/L)
Plasma ultra-sensitive C-reactive protein | 1 year
  Immunoturbidimetric method. Results expressed as milligrams per litre (mg/L)
Plasma vitamin B12 | 1 year
  chemiluminescence immunoassay (CLIA). Results expressed as picograms per millilitre (pg/mL)
Plasma thyroid-stimulating hormone (TSH) | 1 year
  ELISA kit. Values expressed as international micro-units per millilitre (µlU/ml)
Plasma levels of Oleanolic acid | 1 year
  Liquid/liquid extraction and quantification by gas chromatography con flame ionization detection (GC-FID). Values expressed as nanograms per millilitre (ng/mL)
Serum fatty acids composition | 1 year
  Liquid/liquid extraction and quantification by gas chromatography con flame ionization detection (GC-FID). Values expressed as percentage of the total of fatty acids (%)
Plasma adiponectin | 1 year
  ELISA kit. values expressed as picograms per millilitre (pg/mL)
Plasma ceruloplasmin | 1 year
  ELISA kit. values expressed as milligrams per decilitre (mg/dL)
Plasma leptin | 1 year (measures at the time of recruitment and every three months thereafter)
  ELISA kit. values expressed as picograms per millilitre (pg/mL)
Plasma resistin | 1 year
  ELISA kit. values expressed as picograms per millilitre (pg/mL)
Plasma ghrelin | 1 year
  ELISA kit. values expressed as picograms per millilitre (pg/mL)
Plasma catalase | 1 year
  ELISA kit. values expressed as micromole per milligrams of protein (µmol/mg protein)
Plasma superoxide dismutase | 1 year
  ELISA kit. values expressed as units per millilitre (U/mL)
Plasma tumor necrosis factor-alpha (TNF-alpha) | 1 year
  ELISA kit. values expressed as picograms per millilitre (pg/mL)
Plasma interleukine 1-beta | 1 year
  ELISA kit. values expressed as picograms per millilitre (pg/mL)
Plasma interleukine 6 | 1 year
  ELISA kit. values expressed as picograms per millilitre (pg/mL)
Triglycerides in VLDL | 1 year
  the VLDL fraction of plasma lipoproteins will be isolated by ultracentrifugation (230,000 × g for 18 h at 4 0C). Lipds will be extracted by a modification of the Folch's method. Triglycerides are determined by HPLC, and results expressed as milligrams per milligram of protein (mg/mg protein)
Diglycerides in VLDL | 1 year
  the VLDL fraction of plasma lipoproteins will be isolated by ultracentrifugation (230,000 × g for 18 h at 4 0C). Lipds will be extracted by a modification of the Folch's method. Diglycerides are determined by HPLC, and results expressed as milligrams per milligram of protein (mg/mg protein)
Phospholipids in VLDL | 1 year
  the VLDL fraction of plasma lipoproteins will be isolated by ultracentrifugation (230,000 × g for 18 h at 4 0C). Lipds will be extracted by a modification of the Folch's method. Phospholipids are determined by HPLC, and results expressed as milligrams per milligram of protein (mg/mg protein)
Fatty acids composition of VLDL | 1 year
  the VLDL fraction of plasma lipoproteins will be isolated by ultracentrifugation (230,000 × g for 18 h at 4 0C). Lipds will be extracted by a modification of the Folch's method. Fatty acids are derivatized to their methyl esters and analyzed by gas chromatography. The results are expressed as percentage of the total of fatty acids (%)
Apo B in VLDL | 1 year
  Determined by immunoturbidimetry using a commercial kit. Values expressed as micrograms per milligram of protein (µg/mg protein)
Continuous blood glucose monitoring | 1 year
  FreeStyle Libre subcutaneous system (ABBOTT Diagnostics). Values expressed as milligrams per decilitre (mg/dL)
Blood Count - hematocrit | 1 year
  Automated blood analyzer. Results expressed as percentage (%)
Blood Count - red blood cells | 1 year
  Automated blood analyzer. Results expressed as cell count x 10^6 per microlitre (count x 10^6/µL)
Blood Count - hemoglobin | 1 year
  Automated blood analyzer. Results expressed as gram per decilitre (g/dL)
Blood Count - mean corpuscular volume | 1 year
  Automated blood analyzer. Results expressed as femtolitre (fL)
Blood Count - mean corpuscular hemoglobin | 1 year
  Automated blood analyzer. Results expressed as picograms (pg)
Blood Count - leukocytes | 1 year
  Automated blood analyzer. Results expressed as count x 10^3 per microlitre (count x 10^3 /µL)
Blood Count - neutrophils | 1 year
  Automated blood analyzer. Results expressed as count x 10^3 per microlitre (count x 10^3 /µL)
Blood Count - lymphocytes | 1 year
  Automated blood analyzer. Results expressed as count x 10^3 per microlitre (count x 10^3 /µL)
Blood Count - monocytes | 1 year
  Automated blood analyzer. Results expressed as count x 10^3 per microlitre (count x 10^3 /µL)
Blood Count - eosinophils | 1 year
  Automated blood analyzer. Results expressed as count x 10^3 per microlitre (count x 10^3 /µL)
Blood Count - basophils | 1 year
  Automated blood analyzer. Results expressed as count x 10^3 per microlitre (count x 10^3 /µL)
Blood Count - platelets | 1 year
  Automated blood analyzer. Results expressed as count x 10^3 per microlitre (count x 10^3 /µL)
Blood Count - partial thromboplastin time | 1 year
  Automated blood analyzer. Results expressed as seconds (s)
Blood Count - prothrombin time | 1 year
  Automated blood analyzer. Results expressed as seconds (s)
Blood Count - coagulative fibrinogen | 1 year
  Automated blood analyzer. Results expressed as milligrams per decilitre (mg/dL)
Urine pH | 1 year
  Urine pH
Urine density | 1 year
  Automated urine analyzer. Results expressed as milligrams per millilitre (mg/mL)
Glycosuria | 1 year
  Automated urine analyzer. Results expressed as milligrams per decilitre (mg/dL)
Ketone bodies in urine | 1 year
  Automated urine analyzer. Results expressed as millimole per litre (mmol/L)
Presence of nitrite in urine | 1 year
  Automated urine analyzer. Results expressed as negative or positive
Urobilinogen | 1 year
  Automated urine analyzer. Results expressed as milligrams per decilitre (mg/dL)
Urine bilirubin | 1 year
  Automated urine analyzer. Results expressed as milligrams per decilitre (mg/dL)
Urine creatinine | 1 year
  Automated urine analyzer. Results expressed as milligrams per decilitre (mg/dL)
Urine albumin/creatinine ratio (UACR) | 1 year
  Automated urine analyzer. Results expressed as milligrams of albumin per gram of creatinine
Leukocytes in urine | 1 year
  Automated urine analyzer. Results expressed as count x 1 per microlitre (count x 1 /µL)
Presence of sediment in urine | 1 year
  Automated urine analyzer. Results expressed as negative or positive

CONTACTS AND LOCATIONS:
Overall Officials: José María Castellano, PhD, Principal Investigator — Spanish National Research Council (CSIC); Pedro Pablo García-Luna, MD, Principal Investigator — Virgen del Rocío University Hospital
Locations (1):
- Virgen del Rocío University Hospital, Seville, Andalicía, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Castellano JM, Ramos-Romero S, Perona JS. Oleanolic Acid: Extraction, Characterization and Biological Activity. Nutrients. 2022 Jan 31;14(3):623. doi: 10.3390/nu14030623. PMID 35276982
- [Background] Fernandez-Aparicio A, Schmidt-RioValle J, Perona JS, Correa-Rodriguez M, Castellano JM, Gonzalez-Jimenez E. Potential Protective Effect of Oleanolic Acid on the Components of Metabolic Syndrome: A Systematic Review. J Clin Med. 2019 Aug 23;8(9):1294. doi: 10.3390/jcm8091294. PMID 31450844
- [Background] Castellano JM, Guinda A, Delgado T, Rada M, Cayuela JA. Biochemical basis of the antidiabetic activity of oleanolic acid and related pentacyclic triterpenes. Diabetes. 2013 Jun;62(6):1791-9. doi: 10.2337/db12-1215. PMID 23704520
- [Background] Santos-Lozano JM, Rada M, Lapetra J, Guinda A, Jimenez-Rodriguez MC, Cayuela JA, Angel-Lugo A, Vilches-Arenas A, Gomez-Martin AM, Ortega-Calvo M, Castellano JM. Prevention of type 2 diabetes in prediabetic patients by using functional olive oil enriched in oleanolic acid: The PREDIABOLE study, a randomized controlled trial. Diabetes Obes Metab. 2019 Nov;21(11):2526-2534. doi: 10.1111/dom.13838. Epub 2019 Aug 28. PMID 31364228
- See also: website of the OLTRAD Project (BIO-OLTRAD and OLTRAD trials — https://estudiooltrad.wixsite.com/oltrad